CLINICAL TRIAL: NCT04270968
Title: Efficacy of Extracorporeal Shock Wave Therapy (ESWT) on Cervical Myofascial Pain Following Neck Dissection Surgery
Brief Title: Shock Wave Therapy On Cervical Pain Following Neck Dissection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, Department of Physical Therapy, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1857PT
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pain; Cervical Pain
MeSH Terms: conditions — Pain; Neck Pain | interventions — Extracorporeal Shockwave Therapy; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ESWT Group (Experimental): received ESWT once a week for 4 weeks (0.25 ml/mm2, 1000 shocks) plus topical none steroidal anti-inflammatory drug (NSAID; 3 times /day for 4 weeks).
  Interventions: Device: extra-corporeal shock wave therapy
- control group (Experimental): received only topical NSAID.
  Interventions: Drug: topical none steroidal anti-inflammatory drug

INTERVENTIONS:
Device: extra-corporeal shock wave therapy — Extracorporeal Shock Wave Therapy (ESWT) has been introduced efficiently for more than twenty years as a treatment modality in orthopedic and musculoskeletal disorders. ESWT has mechanical and cellular impacts on tissues regeneration and pain management through cavitation bubbles, acoustic micro streaming, and hyper-vascularity that can directly affect tissue calcifications, and modulate cell activity.
  Other Names: shock wave therapy
  Arms: ESWT Group
Drug: topical none steroidal anti-inflammatory drug — participants received 1% topical diclofenac gel on the tender points 3 times /day for 4 weeks.
  Other Names: topical NSAID
  Arms: control group

SUMMARY:
Myofascial pain syndrome (MPS) is a musculoskeletal disorder which is characterized by pain, muscle spasms and muscle tenderness, as well as a limited range of motion, weakness, and rarely, autonomous dysfunction.

DETAILED DESCRIPTION:
The occurrences of morbidity of the neck after cancer therapy were considerable and consisted of neck pain, loss of sensation, and decreased range of motion. Extracorporeal shock wave therapy (ESWT) is one of the treatment options used for patients with myofascial pain syndrome through elimination of ischemia and modulation of vasoneuroactive substance (two major causes of trigger pathophysiology) and mechanical transduction as a cellular response to external stimulation. the aim of this study was to investigate efficacy of extracorporeal shock wave therapy (ESWT) on cervical myofascial pain following neck dissection surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Previous unilateral modified radical neck dissection.
2. Patients with myofascial pain of upper trapezius for at least 3 months.
3. Patients with palpable intramuscular taut band.
4. Restriction in cervical ROM of lateral flexion and rotation.
5. Provocation of the clinical symptoms by compression of the active trigger point

Exclusion Criteria:

1. Patient who received medication or other therapies for MPS within the previous 2 months.
2. Patients with pacemaker, pregnancy
3. Open wound at the treatment area.
4. Cervical myelopathy or radiculopathy, cervical spine fracture or spondylolisthesis.
5. Rheumatoid arthritis.
6. Coagulopathy.
7. Epilepsy or any psychological disorder.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | before treatment
  VAS was utilized for assessing and quantifying pain exhibited by the patients through a 0-10 cm scale. Each subject was informed to mark the line according to the pain intensity experienced at that particular time where '0' means no pain and '10' means worst conceivable pain.
Visual analogue scale | 2 weeks of treatment
  VAS was utilized for assessing and quantifying pain exhibited by the patients through a 0-10 cm scale. Each subject was informed to mark the line according to the pain intensity experienced at that particular time where '0' means no pain and '10' means worst conceivable pain.
Visual analogue scale | after 4 weeks of treatment
  VAS was utilized for assessing and quantifying pain exhibited by the patients through a 0-10 cm scale. Each subject was informed to mark the line according to the pain intensity experienced at that particular time where '0' means no pain and '10' means worst conceivable pain.

SECONDARY OUTCOMES:
Cervical range of motion assessment | before treatment
  Cervical range of motion device (CROM; Performance Attainment Associates) was used for assessment of neck lateral flexion and rotation of both sides. The CROM instrument contains a plastic frame put on the head above the nose and ears, attached at the head back by a Velcro strap to allow precise measure, re-measure and rotational motion in an upright place to avoid individual errors. Two independent inclinometers are connected to the frame and point the head position in relation to the gravity line. Another inclinometer indicates the head position in rotation in relation to a reference position.
Cervical range of motion assessment | 2 weeks of treatment
  Cervical range of motion device (CROM; Performance Attainment Associates) was used for assessment of neck lateral flexion and rotation of both sides. The CROM instrument contains a plastic frame put on the head above the nose and ears, attached at the head back by a Velcro strap to allow precise measure, re-measure and rotational motion in an upright place to avoid individual errors. Two independent inclinometers are connected to the frame and point the head position in relation to the gravity line. Another inclinometer indicates the head position in rotation in relation to a reference position.
Cervical range of motion assessment | after 4 weeks of treatment
  Cervical range of motion device (CROM; Performance Attainment Associates) was used for assessment of neck lateral flexion and rotation of both sides. The CROM instrument contains a plastic frame put on the head above the nose and ears, attached at the head back by a Velcro strap to allow precise measure, re-measure and rotational motion in an upright place to avoid individual errors. Two independent inclinometers are connected to the frame and point the head position in relation to the gravity line. Another inclinometer indicates the head position in rotation in relation to a reference position.

CONTACTS AND LOCATIONS:
Overall Officials: MAGED A BASHA, Dr, Study Director — Assistant Professor, Qassim University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, and figure)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication.
Access Criteria: IPD will be available upon reasonable request by email from the main author after revising the requester qualification relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Result] Guru K, Manoor UK, Supe SS. A comprehensive review of head and neck cancer rehabilitation: physical therapy perspectives. Indian J Palliat Care. 2012 May;18(2):87-97. doi: 10.4103/0973-1075.100820. PMID 23093823
- [Result] Sist T, Miner M, Lema M. Characteristics of postradical neck pain syndrome: a report of 25 cases. J Pain Symptom Manage. 1999 Aug;18(2):95-102. doi: 10.1016/s0885-3924(99)00054-8. PMID 10484856
- [Result] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04270968/Prot_SAP_000.pdf